CLINICAL TRIAL: NCT00736957
Title: A Study of a Long-term Administration of JNS013 in Patients With Chronic Pain
Brief Title: A Long-term Efficacy and Safety Study of Tramadol Hydrochloride Plus Acetaminophen (JNS013) in Japanese Participants With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015115; JNS013-JPN-05
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Acetaminophen; Tramadol; JNS013
MeSH Terms: conditions — Chronic Pain | interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol HCL plus Acetaminophen (Experimental)
  Interventions: Drug: Tramadol Hydrochloride (HCL) plus Acetaminophen (JNS013)

INTERVENTIONS:
Drug: Tramadol Hydrochloride (HCL) plus Acetaminophen (JNS013) — Tramadol hydrochloride 37.5 milligram (mg) plus acetaminophen 325 mg (JNS013) one or two tablets will be given orally four times daily (maximum dose is 8 tablets per day) for 4 weeks during treatment period 1 (restrictions on concomitant treatments will be established) and for 48 weeks during treatment period 2 (permitting modifications to the concomitant drugs/therapies). The dosing interval will be of at least 4 hours.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tramadol hydrochloride plus acetaminophen (JNS013) with long term administration in participants with chronic pain.

DETAILED DESCRIPTION:
This is an open-label (both physician and participant know the name of the study drug), non-randomized, multicenter (when more than one hospital or medical school team work on a medical research study) and long-term efficacy and safety study of JNS013 (combination of tramadol hydrochloride (TRAM) with acetaminophen [APAP]) in participants with chronic pain (aching sensation that persists for more than a few months. It may or may not be associated with trauma or disease, and may persist after the initial injury has healed. Its localization, character, and timing are more vague than with acute pain). This study consists of 4 periods; screening period: 1 week, treatment period I: 4 weeks, treatment period II: 48 weeks and follow-up period: 1 week. During Treatment Period I, restrictions on concomitant treatments will be established and the participants will be treated with one or two tablets of JNS013, four times daily for four weeks. During Treatment Period II, the participants will be treated for 48 weeks using the same dosing method and dose level for JNS013 as was used during Treatment Period I, permitting modifications to the concomitant drugs/therapies as during normal medical care. Throughout both Treatment Period I and Treatment Period II, the decision will be made to permit the participants to select to use either one or two tablets of JNS013 per dose according to the extent of the participant's pain and tolerability. The total duration of treatment period will be of 52 weeks. Efficacy will be assessed using change from baseline in Visual Analogue Scale for pain (VAS24) score at the pre-defined time point until Week 52. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose pain cannot be controlled sufficiently with at least 14-day continuous treatment with identical oral non steroid anti inflammatory drugs (NSAIDs) at a usual maximum dose during 3 months prior to this study
* Ambulatory participants without need for any supportive device or assistance during daily life
* Outpatients
* Participants who do not plan to change the therapeutic policy and content of the medications for underlying disease during screening period to the end of Treatment Period I
* Sustention of chronic pain due to Osteo Arthritis (OA), Low Back Pain (LBP), Rheumatoid Arthritis (RA), Neck Shoulder Arm Syndrome (NSAS), Diabetic Neuropathy (DN), Post herpetic Neuralgia (PHN) or other for at least 3 months

Exclusion Criteria:

* Participants with conditions for which opioids are contraindicated
* Participants with conditions for which APAP are contraindicated
* Participants with history of convulsion or the possibility of convulsive seizure
* Participants with concurrent, previous, or possible alcohol dependence, drug dependence, or narcotic addiction
* Pregnant Participants or those who may be pregnant, lactating mothers, and Participants who wish pregnancy during the study period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (25):
- Japan (25):
  - Chikushi
  - Chūō
  - Fukui
  - Fukuoka
  - Hiratsuka
  - Ichikawa
  - Kashiwa
  - Komatsu
  - Kukichūō
  - Kumamoto
  - Kyoto
  - Mihara
  - Nagoya
  - Nerima City
  - Obihiro
  - Ogi
  - Ohta-Ku
  - Osaka
  - Tagawa
  - Taito-Ku
  - Takaoka
  - Tokyo
  - Urayasu
  - Yame
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 219 participants were enrolled in this study out of which 29 participants did not meet the criteria to transfer to treatment period 1.
Groups:
- Tramadol Hydrochloride Plus Acetaminophen (JNS013): Tramadol hydrochloride 37.5 milligram (mg) plus acetaminophen 325 mg (JNS013) one or two tablets was given orally four times daily (maximum dose was 8 tablets per day) for 4 weeks during treatment period 1 (restrictions on concomitant treatments was established) and for 48 weeks during treatment period 2 (permitting modifications to the concomitant drugs/therapies). The dosing interval was of at least 4 hours.
Period: Overall Study
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Started | 219
Treated | 190
Completed | 97
Not Completed | 122
Not completed — Adverse Event | 43
Not completed — Withdrawal by Subject | 49
Not completed — violation of eligibility criteria | 2
Not completed — did not attend hospital appointments | 1
Not completed — not eligible for Treatment Period I | 22
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] — Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment.
  years | 64.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment.
  Participants
    Female | 106
    Male | 84

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS24) Score at Week 4
Description: Pain over the last 24 hours was assessed by using VAS score ranges from 0 millimeter (mm)=no pain to 100 mm=worst possible pain. An increase in score from baseline represented disease progression and decrease represented improvement.
Time Frame: Baseline and Week 4
Population: Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 190
millimeter
  Baseline | 65.80 (11.629)
  Change at Week 4 | -22.28 (21.189)

2. Primary Outcome: Change From Baseline in VAS24 Score at Week 52
Description: Pain over the last 24 hours was assessed by using VAS score ranges from 0 mm=no pain to 100 mm=worst possible pain. An increase in score from baseline represented disease progression and decrease represented improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 190
millimeter
  Baseline | 65.80 (11.629)
  Change at Week 52 | -36.54 (21.936)

3. Secondary Outcome: Number of Participants With Improvement From Baseline in VAS24 Score
Description: as for outcome 2
Time Frame: Week 4 and 52
Population: Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment. Last Observation Carried Forward (LOCF) method was used.
Measure: Number; unit: participants
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 190
participants
  Improvement of 30 percent or more at Week 4 | 76
  Improvement of 50 percent or more at Week 4 | 51
  Improvement of 30 percent or more at Week 52 | 110
  Improvement of 50 percent or more at Week 52 | 77

4. Secondary Outcome: Pain Intensity Difference (PID) at Week 4
Description: PID is defined as the amount of change in the pain intensity at each evaluation time point (at 2 and 4 hours after the study drug dosing) from the baseline for each participant. Pain Intensity was evaluated on a 4-stage scale ranging from 3=severe pain to 0=no pain. PID ranges from -3 (the worst) to +3 (the most improved).
Time Frame: Week 4
Population: Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment. Participants showing a Pain Intensity (PI) value of 0 prior to dosing at each evaluation time point were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 135
units on a scale
  2 hours after dosing at Week 4 | 0.1 (0.35)
  4 hours after dosing at Week 4 | 0.1 (0.44)

5. Secondary Outcome: Pain Relief (PAR) Score at Week 4
Description: Pain relief was evaluated based on a 5-stage scale from 4 (complete relief) to 0 (no relief). An increase in score represented improvement and decrease represented disease progression
Time Frame: Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 135
units on a scale
  2 hours after dosing at Week 4 | 1.3 (0.91)
  4 hours after dosing at Week 4 | 1.3 (0.99)

6. Secondary Outcome: Pain Relief Combined With Pain Intensity Difference (PRID) at Week 4
Description: PRID was sum of the PID and PAR for each participant at each evaluation time point (2 hours after dosing, 4 hours after dosing). Pain Intensity was evaluated on a 4-stage scale ranges from 3=severe pain to 0=no pain and PID ranges from -3 (the worst) to +3 (the most improved). PAR ranges from 0 (no improved) to +4 (the most improved). PRID ranges from -3 (the worst) to +7 (the most improved).
Time Frame: Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 135
units on scale
  2 hours after dosing at Week 4 | 1.3 (1.06)
  4 hours after dosing at Week 4 | 1.4 (1.20)

7. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Score
Description: SF-36 is a metric for general health and Quality of Life (QOL), consists of 8 sub-scale indices related to health and QOL (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health). Each of the sub-scale scores ranged from 0 to 100, where higher values indicate a better health status or a better mental status.
Time Frame: Baseline, Week 4 and 52
Population: Full analysis set included all participants who met the eligibility criteria, received study medication and had at least one post-treatment efiicacy assessment. 'N' (number of participants analyzed) signifies participants evaluable for this measure and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Number analyzed (Participants) | 190
units on a scale
  Physical functioning:Baseline | 33.7 (17.03)
  Physical functioning:Change at Week 4 (n=150) | 2.9 (9.06)
  Physical functioning:Change at Week 52 (n=96) | 4.1 (12.00)
  Role-physical:Baseline | 35.0 (15.43)
  Role-physical:Change at Week 4 (n=150) | 3.2 (11.51)
  Role-physical:Change at Week 52 (n=96) | 6.0 (13.76)
  Bodily pain:Baseline | 33.7 (6.70)
  Bodily pain:Change at Week 4 (n=150) | 5.5 (7.12)
  Bodily pain:Change at Week 52 (n=96) | 9.0 (8.74)
  General health:Baseline | 42.1 (10.42)
  General health:Change at Week 4 (n=150) | 1.5 (7.74)
  General health:Change at Week 52 (n=96) | 3.9 (8.92)
  Vitality:Baseline | 44.0 (9.82)
  Vitality:Change at Week 4 (n=150) | 2.1 (8.37)
  Vitality:Change at Week 52 (n=96) | 4.9 (9.38)
  Social functioning:Baseline | 41.0 (13.61)
  Social functioning:Change at Week 4 (n=150) | 2.7 (11.36)
  Social functioning:Change at Week 52 (n=96) | 6.0 (11.57)
  Role-emotional:Baseline | 39.4 (14.97)
  Role-emotional:Change at Week 4 (n=150) | 2.6 (12.43)
  Role-emotional:Change at Week 52 (n=96) | 5.2 (14.44)
  Mental health:Baseline | 43.9 (11.50)
  Mental health:Change at Week 4 (n=150) | 2.5 (8.73)
  Mental health:Change at Week 52 (n=96) | 5.5 (10.11)

ADVERSE EVENTS:
Time Frame: From signing of informed consent until study completion (up to 54 weeks)
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen (JNS013)
Serious Adverse Events (participants affected / at risk) | 24/190
Other Adverse Events (participants affected / at risk) | 189/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride Plus Acetaminophen (JNS013) (N=190)
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Cerebral infarction (Nervous system disorders) | 1
Diabetic autonomic nerve neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Sudden deafness (Ear and labyrinth disorders) | 1
Prinzmetal's angina (Cardiac disorders) | 1
Arteriosclerosis obliterans (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Colon polyps (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 1
Upper gastrointestinal tract hemorrhage (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal canal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Ossification of the spinal ligaments (Musculoskeletal and connective tissue disorders) | 1
Ureteral calculus (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Ureteropathy (Renal and urinary disorders) | 1
Fall/tumble (Injury, poisoning and procedural complications) | 1
Open fracture (Injury, poisoning and procedural complications) | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride Plus Acetaminophen (JNS013) (N=190)
Nasopharyngitis (Infections and infestations) | 49
Gastroenteritis (Infections and infestations) | 5
Cystitis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Bronchiectasis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastrointestinal candidiasis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Purulence (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Seasonal allergy (Immune system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 17
Decreased appetite (Metabolism and nutrition disorders) | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 15
Delusion (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Listless (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Affect lability (Psychiatric disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 52
Somnolence (Nervous system disorders) | 38
Headache (Nervous system disorders) | 28
Dysgeusia (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 4
Cervicobrachial syndrome (Nervous system disorders) | 3
Carpal tunnel syndrome (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
IVth nerve paralysis (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Occipital neuralgia (Nervous system disorders) | 1
Conjunctivitis allergic (Eye disorders) | 4
Conjunctival haemorrhage (Eye disorders) | 2
Diabetic retinopathy (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Posterior capsule opacification (Eye disorders) | 1
Vitreous detachment (Eye disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 2
Deafness neurosensory (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Palpitations (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 14
Hot flush (Vascular disorders) | 4
Blood pressure fluctuation (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Arteriosclerosis obliterans (Vascular disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 101
Constipation (Gastrointestinal disorders) | 75
Vomiting (Gastrointestinal disorders) | 68
Stomach discomfort (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 16
Gastritis (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 6
Reflux oesophagitis (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 3
Periodontitis (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Melanosis coli (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1
Oral mucosa erosion (Gastrointestinal disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11
Eczema (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5
Cold sweat (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Senile pruritus (Skin and subcutaneous tissue disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 1
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 7
Haematuria (Renal and urinary disorders) | 1
Micturition disorder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Malaise (General disorders) | 15
Feeling abnormal (General disorders) | 13
Thirst (General disorders) | 12
Pyrexia (General disorders) | 8
Oedema peripheral (General disorders) | 7
Chest discomfort (General disorders) | 3
Oedema (General disorders) | 2
Application site dermatitis (General disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Feeling cold (General disorders) | 1
Injection site haematoma (General disorders) | 1
Pain (General disorders) | 1
Peripheral coldness (General disorders) | 1
Vessel puncture site haematoma (General disorders) | 1
Weight decreased (Investigations) | 23
Gamma-glutamyltransferase increased (Investigations) | 21
Blood creatine phosphokinase increased (Investigations) | 19
Blood triglycerides increased (Investigations) | 14
Blood pressure increased (Investigations) | 11
Blood urea increased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 9
Glucose urine present (Investigations) | 7
Blood urine present (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 6
Blood potassium increased (Investigations) | 5
Liver function test abnormal (Investigations) | 5
Eosinophil percentage increased (Investigations) | 5
White blood cell count increased (Investigations) | 4
Haemoglobin decreased (Investigations) | 3
Weight increased (Investigations) | 3
Protein urine present (Investigations) | 3
Albumin urine present (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood pressure systolic increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Red blood cell count decreased (Investigations) | 2
Platelet count increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure diastolic decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Neutrophil percentage decreased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 11
Wound (Injury, poisoning and procedural complications) | 5
Excoriation (Injury, poisoning and procedural complications) | 3
Thermal burn (Injury, poisoning and procedural complications) | 3
Joint sprain (Injury, poisoning and procedural complications) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Blood lactate dehydrogenase increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.